CLINICAL TRIAL: NCT02592395
Title: Phase I Study of FOLFIRINOX Electrochemotherapy in the Treatment of Pancreatic Adenocarcinoma
Brief Title: Study of FOLFIRINOX Electrochemotherapy in the Treatment of Pancreatic Adenocarcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI transferred to another institution and did not take this study with him.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-15-0659
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: pancreatic adenocarcinoma; electrochemotherapy; electroporation; radiogenomics; imaging; magnetic resonance spectroscopy
MeSH Terms: interventions — folfirinox; Electroporation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Electrochemotherapy with FOLFIRINOX (Experimental): During the first cycle of chemotherapy, patients will receive electroporation of the primary pancreatic tumor prior to administration of chemotherapy with FOLFIRINOX . The schedule of administration of FOLFIRINOX will be administered as per standard of care.
  Interventions: Drug: FOLFIRINOX; Device: Electroporation

INTERVENTIONS:
Drug: FOLFIRINOX — The chemotherapy schedule will include administration of FOLFIRINOX (5-Fluorouracil, Irinotecan, Oxaliplatin, and Leucovorin) will be:
  Day 1: Oxaliplatin at 85mg/m2 over 120 minutes, Irinotecan 180mg/m2 over 90 minutes, Leucovorin 400mg/m2 over 90minutes, 5-Fluorouracil (5-FU) 1200mg/m2/day continuous infusion (CIV) over 46 hours. Day 3: 5-FU CIV pump will be disconnected. Neulasta injection 6mg subcutaneous
Device: Electroporation — Irreversible electroporation (IRE) will be performed under computed tomography (CT) guidance, during which 2 to 6 needles are advanced into the pancreatic tumor where a specified field strength will be applied.
  Other Names: Irreversible electroporation (IRE)

SUMMARY:
The purpose of this study is to see how well electrochemotherapy works at treating people with Stage III pancreatic adenocarcinoma. Electrochemotherapy is a treatment that combines electroporation and chemotherapy administration. Electroporation uses an electric current to produce holes in pancreatic tumor, which causes the tumor cells to die or take up a higher concentration of administered chemotherapy agent. This study will test the safety and look at the effect of electrochemotherapy in the treatment of stage III pancreatic adenocarcinoma. This study will also help to find the safest and most effective amount of electroporation voltage to apply to this type of tumor.

DETAILED DESCRIPTION:
This is a phase I dose escalation trial using a 3 + 3 dose escalation scheme to evaluate the maximum tolerated field strength dose of administered irreversible electroporation in combination with chemotherapy. During the first cycle of chemotherapy, patients will receive electroporation of the primary pancreatic tumor prior to administration of chemotherapy with FOLFIRINOX. The schedule of administration of FOLFIRINOX will be administered as per standard of care. The investigators will use non-invasive dynamic magnetic resonance imaging and magnetic resonance spectroscopy to detect and describe changes within the tumor. Safety will be determined by assessing the number of class three or higher toxicity events in cohorts of 6 patients at progressively higher electroporation voltages. The maximum tolerated dose (MTD) will be defined as one voltage level less than the voltage at which two or more patients out of six total patients have a class three or higher toxicity event.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven pancreatic carcinoma which is safely accessible by percutaneous methods;
* Locally advanced un-resectable pancreatic adenocarcinoma;
* At least one measurable lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria (longest diameter >=20 mm using conventional techniques or >=10 mm with spiral CT or MRI scan);
* WHO performance status (PS) < 2 or Eastern Cooperative Oncology Group < 2;
* Age >18;
* Life expectancy > 3 months;
* No history of gastric or esophageal varices;
* No active, uncontrolled infection;
* All patients must have adequate physiologic (hematologic, renal and hepatic) reserves as evidenced by: neutrophil count >1500/mL; platelet count >100,000/mL; serum creatinine <1.5x the upper limit of normal (ULN) value; serum glutamic-pyruvic transaminase (SGPT) <2.5 x ULN and bilirubin <1.5 x ULN functions
* Pain and biliary obstruction controlled before the start of the study
* Absence of psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule;
* Women of childbearing potential (defined as sexually mature woman who 1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or 2) has not been naturally post-menopausal for at last 24 consecutive months) must have a negative pregnancy test prior to starting therapy. Men and women of childbearing potential must be willing to use effective contraceptive while on treatment and for a reasonable period thereafter.

Exclusion Criteria:

* Prior chemotherapy with FOLFIRINOX;
* Prior history of pancreatic electroporation;
* Untreatable contrast allergy;
* History of allergy or hypersensitivity to gemcitabine, nab-paclitaxel, or any of the excipients;
* Presence of metal biliary stent;
* Psychosis or seizures;
* Evidence of serious gastrointestinal bleeding or bowel obstruction;
* Pregnant or lactating women;
* Women of childbearing potential who are not using adequate protection;
* Inability to tolerate MRI imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experienced dose limiting toxicities (DLTs) | 4 weeks
  A dose limiting toxicity (DLT) is any Grade 3 or 4 adverse event (AE) using the Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE 4.0) that is possibly related to the electrochemotherapy treatment. CTCAE 4.0 Grade 3 is a severe AE and Grade 4 is a life-threatening or disabling AE. DLTs are collected to determine the Maximum Tolerated Dose (MTD), which is defined as as one field strength level less than the field strength at which two or more patients out of six total patients experience a DLT.

SECONDARY OUTCOMES:
Number of participants who demonstrated no clinical change or clinical improvement in pancreatic adenocarcinoma outcome as assessed by time to progression | 1 year
  Time to progression is the time after treatment until tumor enlargement or metastatic disease is identified.
Number of participants who demonstrated no clinical change or clinical improvement in pancreatic adenocarcinoma outcome as assessed by one year survival | 1 year
  One year survival is the number of patients who are alive one year after treatment.
Number of participants who demonstrated no clinical change or clinical improvement in pancreatic adenocarcinoma outcome as assessed by tumor imaging | 1 year
  We will assess tumor size changes and tumor staging through magnetic resonance imaging (MRI).
Number of participants who demonstrated diffusion weighted magnetic resonance imaging (MRI) changes | 1 year
Number of participants who demonstrated magnetic resonance spectroscopy (MRS) changes | 1 year
Number of groups of patients who have similar pancreatic tumor gene expression characteristics after electrochemotherapy | 1 year
  Gene expression characteristics are identified by biopsy specimen evaluation.
Number of groups of patients who have similar imaging characteristics after electrochemotherapy | 1 year
  Imaging characteristics are evaluated by MRI and MRS.
Number of groups of patients who have similar clinical outcomes after electrochemotherapy | 1 year
  Clinical outcomes are evaluated by time to progression and 1 year survival. Time to progression is the time after treatment until tumor enlargement or metastatic disease is identified. One year survival is the number of patients who are alive one year after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Derek L West, MD, MS, Principal Investigator — The University of Texas Health Science Center, Houston